CLINICAL TRIAL: NCT01846273
Title: A 24-month, Phase IV, Randomized, Double Masked, Multi-center Study of Ranibizumab Monotherapy or Ranibizumab in Combination With Verteporfin Photodynamic Therapy on Visual Outcome in Patients With Symptomatic Macular Polypoidal Choroidal Vasculopathy
Brief Title: Visual Outcome in Patients With Symptomatic Macular Polypoidal Choroidal Vasculopathy (PCV) Treated With Either Ranibizumab as Monotherapy or Combined With Verteporfin Photodynamic Therapy (vPDT)
Acronym: EVEREST II
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CRFB002A2412
Record Dates: First submitted 2013-04-29; First posted 2013-05-03 (Estimated); Results first posted 2019-06-07 (Actual); Last update posted 2019-06-07 (Actual); Status verified 2019-03

CONDITIONS: Age-related Macular Degeneration; Polypoidal Choroidal Vasculopathy
Keywords: Polypoidal choroidal vasculopathy; Visual acuity; Ranibizumab; Verteporfin PDT
MeSH Terms: conditions — Macular Degeneration; Polypoidal Choroidal Vasculopathy | interventions — Ranibizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ranibizumab + vPDT (Experimental): Treatment initiation with Ranibizumab and verteporfin PDT (vPDT), with re-treatment need (either Ranibizumab alone or combined with vPDT) determined at monthly visits based on defined retreatment criteria
  Interventions: Drug: Ranibizumab; Drug: Verteporfin PDT
- Ranibizumab monotherapy (Active Comparator): Treatment initiation with Ranibizumab and Sham PDT, with re-treatment need (either Ranibizumab alone or combined with Sham PDT) determined at monthly visits based on defined retreatment criteria
  Interventions: Drug: Ranibizumab; Drug: Sham PDT

INTERVENTIONS:
Drug: Ranibizumab — Intravitreal injection of 0.5 mg ranibizumab
  Other Names: Lucentis
Drug: Verteporfin PDT — Infusion of 30 ml verteporfin in 5% dextrose solution followed by 83 sec of laser light (50J/cm2; 600mW/cm2; 689 nm)
  Arms: Ranibizumab + vPDT
Drug: Sham PDT — Infusion of 30 ml 5% dextrose solution followed by 83 sec of laser light (50J/cm2; 600mW/cm2; 689 nm)
  Arms: Ranibizumab monotherapy

SUMMARY:
This study compared the effect of ranibizumab administered as monotherapy versus ranibizumab administered in combination with verteporfin photodynamic therapy (PDT) on visual acuity in patients with symptomatic macular polypoidal choroidal vasculopathy (PCV). The results of this study provided long-term safety and efficacy data used to generate further guidance on the management of patients with PCV.

DETAILED DESCRIPTION:
Patients were randomized to the study in 2 treatment groups: ranibizumab + vPDT combination therapy, and ranibizumab monotherapy. Based on the results of the primary analysis at Month 12, patients still in the ranibizumab monotherapy group at the time of the switch cut-off time point were switched to the ranibizumab + vPDT combination therapy group until study exit. A total of 168 and 154 patients were included in the ranibizumab + vPDT combined therapy and ranibizumab monotherapy groups, respectively for the FAS (Month 12 analysis). However, the safety set included 172 and 149 patients, respectively. Four patients in the combination therapy group never took vPDT . Among them, 1 patient actually received verteporfin injection but no laser injection. Thus a total of 3 patients (4-1) in the combination therapy group did not take the actual full vPDT treatment. Additionally, 7 patients in the monotherapy group received vPDT and 1 patient from the monotherapy group did not receive ranibizumab treatment. Considering the above numbers, safety set included 172 patients (i.e., 168-3+7) in the ranibizumab + vPDT combination therapy group and 149 patients (i.e., 154-7+3-1) in the ranibizumab monotherapy group for Month 12 analysis. For the Month 24 safety analysis, the 14 patients in the ranibizumab monotherapy group who were switched to ranibizumab +vPDT combination therapy group were analyzed as a separate group, ie, ranibizumab 0.5 mg + vPDT (switched).

.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of symptomatic macular PCV in the study eye
* A qualifying vision score at study entry
* A qualifying lesion size in the study eye at study entry

Exclusion Criteria:

* Active inflammation or infection in the study eye
* Uncontrolled intraocular pressure in the stuy eye
* Ocular condition in the study eye which may impact vision and confound study outcomes
* Prior treatment of the study eye with anti-VEGF therapy, verteporfin PDT, other laser and surgical interventions, intraocular corticosteroids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 321 (Actual)
Dates: Start 2013-08-07 (Actual); Primary Completion 2016-03-11 (Actual); Study Completion 2017-03-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (34):
- Novartis Investigative Site, Hong Kong, Hong Kong
- Japan (19):
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Fukuoka, Fukuoka
  - Novartis Investigative Site, Fukushima, Fukushima
  - Novartis Investigative Site, Maebashi, Gunma
  - Novartis Investigative Site, Amagasaki, Hyōgo
  - Novartis Investigative Site, Kobe, Hyōgo
  - Novartis Investigative Site, Inashiki-gun, Ibaraki
  - Novartis Investigative Site, Kita-gun, Kagawa-ken
  - Novartis Investigative Site, Sakyo-ku, Kyoto
  - Novartis Investigative Site, Tsu, Mie-ken
  - Novartis Investigative Site, Okayama, Okayama-ken
  - Novartis Investigative Site, Hirakata, Osaka
  - Novartis Investigative Site, Osaka, Osaka
  - Novartis Investigative Site, Ohtsu-city, Shiga
  - Novartis Investigative Site, Bunkyo Ku, Tokyo
  - Novartis Investigative Site, Chiyoda-ku, Tokyo
  - Novartis Investigative Site, Mitaka, Tokyo
  - Novartis Investigative Site, Shinjuku Ku, Tokyo
  - Novartis Investigative Site, Chiba
- Malaysia (2):
  - Novartis Investigative Site, Batu Caves, Selangor
  - Novartis Investigative Site, Petaling Jaya, Selangor
- Novartis Investigative Site, Singapore, Singapore
- South Korea (4):
  - Novartis Investigative Site, Seongnam-si, Gyeonggi-do
  - Novartis Investigative Site, Seoul, Korea
  - Novartis Investigative Site, Seoul, Seocho-gu
  - Novartis Investigative Site, Seoul
- Taiwan (5):
  - Novartis Investigative Site, Taipei, Taiwan, ROC
  - Novartis Investigative Site, Changhua
  - Novartis Investigative Site, Kaohsiung City
  - Novartis Investigative Site, Taipei
  - Novartis Investigative Site, Taoyuan District
- Thailand (2):
  - Novartis Investigative Site, Songkhla, Hat Yai
  - Novartis Investigative Site, Bangkok

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yanagi Y, Mori R, Teo KYC, Park KH, Ngah NF, Chen SJ, Ruamviboonsuk P, Kondo N, Lee WK, Rajagopalan R, Obata R, Wong IYH, Chee C, Terasaki H, Sekiryu T, Chen SC, Lai TYY, Cheung G, Honda S. Six-year findings of polypoidal choroidal vasculopathy in the EVEREST II study: Japanese subgroup analysis. Jpn J Ophthalmol. 2025 Nov;69(6):894-901. doi: 10.1007/s10384-025-01228-w. Epub 2025 Jun 12. PMID 40504425
- [Derived] Teo KYC, Park KH, Ngah NF, Chen SJ, Ruamviboonsuk P, Mori R, Kondo N, Lee WK, Rajagopalan R, Obata R, Wong IYH, Chee C, Terasaki H, Sekiryu T, Chen SC, Yanagi Y, Honda S, Lai TYY, Cheung CMG. Six-Year Outcomes in Subjects with Polypoidal Choroidal Vasculopathy in the EVEREST II Study. Ophthalmol Ther. 2024 Apr;13(4):935-954. doi: 10.1007/s40123-024-00888-0. Epub 2024 Feb 3. PMID 38308746
- [Derived] Lim TH, Lai TYY, Takahashi K, Wong TY, Chen LJ, Ruamviboonsuk P, Tan CS, Lee WK, Cheung CMG, Ngah NF, Patalauskaite R, Margaron P, Koh A; EVEREST II Study Group. Comparison of Ranibizumab With or Without Verteporfin Photodynamic Therapy for Polypoidal Choroidal Vasculopathy: The EVEREST II Randomized Clinical Trial. JAMA Ophthalmol. 2020 Sep 1;138(9):935-942. doi: 10.1001/jamaophthalmol.2020.2443. PMID 32672800
- [Derived] Koh A, Lai TYY, Takahashi K, Wong TY, Chen LJ, Ruamviboonsuk P, Tan CS, Feller C, Margaron P, Lim TH, Lee WK; EVEREST II study group. Efficacy and Safety of Ranibizumab With or Without Verteporfin Photodynamic Therapy for Polypoidal Choroidal Vasculopathy: A Randomized Clinical Trial. JAMA Ophthalmol. 2017 Nov 1;135(11):1206-1213. doi: 10.1001/jamaophthalmol.2017.4030. PMID 28983556

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted in the following jurisdictions: Japan (25 centers), Malaysia (2 centers), Singapore (4 centers), Hong Kong (2 centers), Taiwan (6 centers), Thailand (3 centers) and Korea (5 centers).
Pre-assignment Details: The enrollment number in the protocol section reflects the number of participants treated (321). The total number in the participant flow and baseline characteristics sections reflects the number of participants randomized (322).
Groups:
- Ranibizumab 0.5 mg + vPDT: Treatment initiation with Ranibizumab and verteporfin PDT (vPDT), with re-treatment need (either Ranibizumab alone or combined with vPDT)
- Ranibizumab 0.5 mg: Treatment initiation with Ranibizumab and Sham PDT, with re-treatment need (either Ranibizumab alone or combined with Sham PDT)
- Ranibizumab 0.5 mg + vPDT (Switched): Based on the results of the primary analysis at Month 12, patients still in the Ranibizumab monotherapy group (Ranibizumab 0.5 mg) at the time of the switch cut-off time point were switched to the ranibizumab + vPDT combination therapy group until study exit
Period: Overall Study
Arm/Group | Ranibizumab 0.5 mg + vPDT | Ranibizumab 0.5 mg | Ranibizumab 0.5 mg + vPDT (Switched)
Started (Full Analysis Set) | 168 | 113 | 41
Safety Analysis Set | 172 | 135 | 14
Completed | 146 | 87 | 41
Not Completed | 22 | 26 | 0
Not completed — Adverse Event | 9 | 7 | 0
Not completed — Subject withdrew consent | 5 | 8 | 0
Not completed — Lost to Follow-up | 2 | 1 | 0
Not completed — Administrative problems | 1 | 0 | 0
Not completed — Death | 2 | 1 | 0
Not completed — Disease Progression | 0 | 4 | 0
Not completed — Protocol Deviation | 2 | 3 | 0
Not completed — Physician Decision | 1 | 2 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set
Groups:
- Total: Total of all reporting groups
Arm/Group | Ranibizumab 0.5 mg + vPDT | Ranibizumab 0.5 mg | Ranibizumab 0.5 mg + vPDT (Switched) | Total
Number analyzed (Participants) | 168 | 113 | 41 | 322
Age, Continuous [Mean (Standard Deviation); unit: years] | 68 (8.54) | 67.8 (9.19) | 69.2 (8.57) | 68.1 (8.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59 | 30 | 8 | 97
  Male | 109 | 83 | 33 | 225

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Best Corrected Visual Acuity (BCVA) at Month 12 - Study Eye
Description: Best Corrected Visual Acuity (BCVA) was assessed during all study visits using best correction determined from protocol refraction at a starting test distance of 4 meters. VA measurements were taken in a sitting position using Early Treatment Diabetic Retinopathy Study (ETDRS)-like visual acuity testing charts. The BCVA score is the number of letters read correctly by the patient, hence an increase in score indicates improvement in acuity.
Time Frame: Baseline, Month 12
Population: Full Analysis Set (FAS) using the Last Observation Carried Forward (LOCF) approach for imputing missing data
Measure: Least Squares Mean (Standard Error); unit: Letters
Arm/Group | Ranibizumab 0.5 mg + vPDT | Ranibizumab 0.5 mg
Number analyzed (Participants) | 168 | 154
Letters | 8.3 (1.00) | 5.1 (1.06)
Statistical Analysis 1: Comparison: Ranibizumab 0.5 mg + vPDT vs Ranibizumab 0.5 mg; Test type: Non-Inferiority — pre-defined non-inferiority margin of 5 letters; p < 0.001, ANCOVA; Least Squares Mean = 3.2, 95% CI 1-sided [lower limit 0.38]

2. Primary Outcome: Number of Patients With Complete Polyp Regression From Baseline at Month 12 - Study Eye
Description: Polyp regression was based on the Indocyanine green angiography (ICGA) assessment by the Central Reading Center (CRC). A patient was considered to have complete polyp regression if the presence of polyps, as assessed by CRC, had value "No." Polyp regression which may lead to disease stabilization and consequently better vision.
Time Frame: Baseline, Month 12
Population: Full Analysis Set (FAS) using the Last Observation Carried Forward (LOCF) approach for imputing missing data
Measure: Number; unit: Participants
Arm/Group | Ranibizumab 0.5 mg + vPDT | Ranibizumab 0.5 mg
Number analyzed (Participants) | 168 | 154
Participants | 115 | 52
Statistical Analysis 1: Comparison: Ranibizumab 0.5 mg + vPDT vs Ranibizumab 0.5 mg; Test type: Superiority; p < 0.0001, Fisher Exact

3. Secondary Outcome: Mean Change From Baseline in Best-Corrected Visual Acuity (BCVA) at Month 24 - Study Eye
Description: Best Corrected Visual Acuity (BCVA) was assessed during all study visits using best correction determined from protocol refraction at a starting test distance of 4 meters. VA measurements were taken in a sitting position using Early Treatment Diabetic Retinopathy Study (ETDRS)-like visual acuity testing charts at a starting test distance of 4 meters. The BCVA score is the number of letters read correctly by the patient, hence an increase in score indicates improvement in acuity.
Time Frame: Baseline, Month 24
Population: All patients with a BCVA value for both baseline and Month 24
Measure: Least Squares Mean (Standard Error); unit: Letters
Arm/Group | Ranibizumab 0.5 mg + vPDT | Ranibizumab 0.5 mg | Ranibizumab 0.5 mg + vPDT (Switched)
Number analyzed (Participants) | 168 | 113 | 41
Letters | 9.7 (11.74) | 5.4 (12.75) | 6.1 (13.84)

4. Secondary Outcome: Percentage of Patients With BCVA (Letters) Change From Baseline at Month 24 - Study Eye
Description: BCVA score was based on the number of letters read correctly on the Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity chart assessed at a starting distance of 4 meters. An ETDRS visual acuity score of 85 is approximately 20/20.
Time Frame: Baseline, Month 24
Population: All participants with a BCVA value for both Baseline and Month 24.
Measure: Number; unit: Percentage of participants
Arm/Group | Ranibizumab 0.5 mg + vPDT | Ranibizumab 0.5 mg | Ranibizumab 0.5 mg + vPDT (Switched)
Number analyzed (Participants) | 168 | 113 | 41
Percentage of participants
  ≥ 5 letters gain: number analyzed (Participants) | 146 | 87 | 41
  ≥ 5 letters gain | 74.0 | 57.5 | 51.2
  ≥ 10 letters gain: number analyzed (Participants) | 146 | 87 | 41
  ≥ 10 letters gain | 51.4 | 36.8 | 43.9
  ≥ 15 letters gain: number analyzed (Participants) | 146 | 87 | 41
  ≥ 15 letters gain | 30.8 | 24.1 | 24.4
  < 5 letters loss: number analyzed (Participants) | 131 | 74 | 34
  < 5 letters loss | 89.7 | 85.1 | 82.9
  < 10 letters loss: number analyzed (Participants) | 138 | 80 | 37
  < 10 letters loss | 94.5 | 92.0 | 90.2
  < 15 letters loss: number analyzed (Participants) | 139 | 83 | 38
  < 15 letters loss | 95.2 | 95.4 | 92.7
  < 30 letters loss: number analyzed (Participants) | 145 | 85 | 41
  < 30 letters loss | 99.3 | 97.7 | 100

5. Secondary Outcome: Maintenance of BCVA (Within 5 Letter Change) at Month 12 and 24 Compared to BCVA at the Time Point of First Ranibizumab Treatment Interruption
Description: Best Corrected Visual Acuity (BCVA) was assessed using best correction determined from protocol refraction at a starting test distance of 4 meters. VA measurements were taken in a sitting position using Early Treatment Diabetic Retinopathy Study (ETDRS)-like visual acuity testing charts at a starting test distance of 4 meters.
Time Frame: Month 3, Month 12, Month 24
Population: Prior to DB lock, the statistical analysis plan was amended and this endpoint was removed (initially included in order to assess VA maintenance during the PRN phase after the loading phase of ranibizumab 0.5 mg). When SAP was finalized, this question had already been addressed (CRF002A2413 (NCT01775124), FVF4579g (NCT00891735)): no data collected.
Arm/Group | Ranibizumab 0.5 mg + vPDT | Ranibizumab 0.5 mg | Ranibizumab 0.5 mg + vPDT (Switched)
Number analyzed (Participants) | 0 | 0 | 0

6. Secondary Outcome: Change in BCVA at Month 12 and 24 Compared to the Time Point of First Ranibizumab Treatment Interruption
Description: as for outcome 5
Time Frame: Month 3, Month 12, Month 24
Population: as for outcome 5
Arm/Group | Ranibizumab 0.5 mg + vPDT | Ranibizumab 0.5 mg | Ranibizumab 0.5 mg + vPDT (Switched)
Number analyzed (Participants) | 0 | 0 | 0

7. Secondary Outcome: Percentage of Patients With Complete Polyp Regression at Months 6 and 24 - Study Eye
Description: as for outcome 2
Time Frame: Month 6, Month 24
Population: All patients who attended the specific visit
Measure: Number; unit: Percentage of participants
Arm/Group | Ranibizumab 0.5 mg + vPDT | Ranibizumab 0.5 mg | Ranibizumab 0.5 mg + vPDT (Switched)
Number analyzed (Participants) | 168 | 113 | 41
Percentage of participants
  Month 6 - Total: number analyzed (Participants) | 157 | 102 | 41
  Month 6 - Total | 100 | 100 | 100
  Month 6 - Yes: number analyzed (Participants) | 112 | 31 | 9
  Month 6 - Yes | 71.3 | 30.4 | 22.0
  Month 6 - No: number analyzed (Participants) | 45 | 71 | 32
  Month 6 - No | 28.7 | 69.6 | 78.0
  Month 6 - Can't grade: number analyzed (Participants) | 0 | 0 | 0
  Month 24 - Total: number analyzed (Participants) | 143 | 86 | 40
  Month 24 - Total | 100 | 100 | 100
  Month 24 - Yes: number analyzed (Participants) | 81 | 23 | 19
  Month 24 - Yes | 56.6 | 26.7 | 47.5
  Month 24 - No: number analyzed (Participants) | 62 | 63 | 21
  Month 24 - No | 43.4 | 73.3 | 52.5
  Month 24 - Can't grade: number analyzed (Participants) | 0 | 0 | 0

8. Secondary Outcome: Percentage of Patients With Presence of Leakage at Month 6, Month 12 and Month 24 - Study Eye
Description: Presence of lesion leakage was based on Fluorescein Angiography (FA) as assessed by the Central Reading Center (CRC). The presence of leakage may lead to disease progression and worsening vision.
Time Frame: Month 6, Month 12 and Month 24
Population: All patients who attended the specific visit
Measure: Number; unit: Percentage of participants
Arm/Group | Ranibizumab 0.5 mg + vPDT | Ranibizumab 0.5 mg | Ranibizumab 0.5 mg + vPDT (Switched)
Number analyzed (Participants) | 168 | 113 | 41
Percentage of participants
  Month 6 - Total: number analyzed (Participants) | 158 | 102 | 41
  Month 6 - Total | 100 | 100 | 100
  Month 6 - Yes: number analyzed (Participants) | 68 | 75 | 32
  Month 6 - Yes | 43 | 73.5 | 78
  Month 6 - No: number analyzed (Participants) | 87 | 27 | 22
  Month 6 - No | 55.1 | 26.5 | 22
  Month 6 - Can't grade: number analyzed (Participants) | 1 | 0 | 0
  Month 6 - Can't grade | 0.6 |  |
  Month 6 - Missing: number analyzed (Participants) | 2 | 0 | 0
  Month 6 - Missing | 1.3 |  |
  Month 12 - Total: number analyzed (Participants) | 155 | 95 | 41
  Month 12 - Total | 100 | 100 | 100
  Month 12 - Yes: number analyzed (Participants) | 74 | 69 | 33
  Month 12 - Yes | 47.7 | 72.6 | 80.5
  Month 12 - No: number analyzed (Participants) | 80 | 26 | 8
  Month 12 - No | 51.6 | 27.4 | 19.5
  Month 12 - Can't grade: number analyzed (Participants) | 0 | 0 | 0
  Month 12 - Missing: number analyzed (Participants) | 1 | 0 | 0
  Month 12 - Missing | 0 |  |
  Month 24 - Total: number analyzed (Participants) | 146 | 86 | 41
  Month 24 - Total | 100 | 100 | 100
  Month 24 - Yes: number analyzed (Participants) | 83 | 56 | 23
  Month 24 - Yes | 56.8 | 65.1 | 56.1
  Month 24 - No: number analyzed (Participants) | 59 | 30 | 16
  Month 24 - No | 40.4 | 34.9 | 39
  Month 24 - Can't grade: number analyzed (Participants) | 1 | 0 | 1
  Month 24 - Can't grade | 0.7 |  | 2.4
  Month 24 - Missing: number analyzed (Participants) | 3 | 0 | 1
  Month 24 - Missing | 2.1 |  | 2.4

9. Secondary Outcome: Mean Change From Baseline in Investigator-Assessed Central Subfield Retinal Thickness (CSFT) at Month 24 - Study Eye
Description: The thickness of the retina was measured using Spectral Domain (SD) optical coherence tomography (OCT) equipment (SD-OCT) and reported as a difference, in micrometers. A negative number indicates a reduction in thickness, whereas a positive number indicates an increase. An increase in thickness may indicate a progression of the underlying disease.
Time Frame: Baseline, Month 24
Population: All patients with a value at baseline and at Month 24
Measure: Least Squares Mean (Standard Error); unit: Micrometers
Arm/Group | Ranibizumab 0.5 mg + vPDT | Ranibizumab 0.5 mg | Ranibizumab 0.5 mg + vPDT (Switched)
Number analyzed (Participants) | 168 | 113 | 41
Micrometers
  Value at Baseline: number analyzed (Participants) | 146 | 87 | 41
  Value at Baseline | 401.6 (142.74) | 390 (124.12) | 412.5 (143.16)
  Value at Month 24: number analyzed (Participants) | 146 | 87 | 41
  Value at Month 24 | 248.8 (64.7) | 294.5 (108.61) | 273.8 (73.31)
  Change from Baseline: number analyzed (Participants) | 146 | 87 | 41
  Change from Baseline | -152.9 (129.74) | -95.5 (148.36) | -138.7 (124.94)

10. Secondary Outcome: Total Number of Ranibizumab Injections Received in the Study Eye Prior to Month 12
Time Frame: Baseline, Month 12
Population: Safety Analysis Set
Measure: Number; unit: injections
Arm/Group | Ranibizumab 0.5 mg + vPDT | Ranibizumab 0.5 mg
Number analyzed (Participants) | 172 | 149
injections | 887 | 1089

11. Secondary Outcome: Total Number of Verteporfin/Sham PDT Injections Received in the Study Eye Prior to Month 12
Time Frame: Baseline, Month 12
Population: Safety Analysis Set
Measure: Number; unit: injections
Arm/Group | Ranibizumab 0.5 mg + vPDT | Ranibizumab 0.5 mg
Number analyzed (Participants) | 172 | 149
injections | 264 | 345

12. Secondary Outcome: Total Number of Ranibizumab Injections Received in the Study Eye Prior to Month 24
Time Frame: Baseline, Month 24
Population: Safety Analysis Set
Measure: Number; unit: injections
Arm/Group | Ranibizumab 0.5 mg + vPDT | Ranibizumab 0.5 mg | Ranibizumab 0.5 mg + vPDT (Switched)
Number analyzed (Participants) | 172 | 135 | 14
injections | 1422 | 1625 | 225

13. Secondary Outcome: Total Number of Verteporfin/Sham PDT Injections Received in the Study Eye Prior to Month 24
Time Frame: Baseline, Month 24
Population: Safety Analysis Set
Measure: Number; unit: injections
Arm/Group | Ranibizumab 0.5 mg + vPDT | Ranibizumab 0.5 mg | Ranibizumab 0.5 mg + vPDT (Switched)
Number analyzed (Participants) | 172 | 135 | 14
injections | 389 | 459 | 81

14. Secondary Outcome: Total Number of Ranibizumab Injections Received in the Study Eye From Month 3 to Month 12
Time Frame: Month 3, Month 12
Population: Safety Analysis Set
Measure: Number; unit: injections
Arm/Group | Ranibizumab 0.5 mg + vPDT | Ranibizumab 0.5 mg
Number analyzed (Participants) | 172 | 149
injections | 378 | 651

15. Secondary Outcome: Total Number of Ranibizumab Injections Received in the Study Eye From Month 3 to Month 24
Time Frame: Month 3, Month 24
Population: Safety Analysis Set
Measure: Number; unit: injections
Arm/Group | Ranibizumab 0.5 mg + vPDT | Ranibizumab 0.5 mg | Ranibizumab 0.5 mg + vPDT (Switched)
Number analyzed (Participants) | 172 | 135 | 14
injections | 913 | 1229 | 183

16. Secondary Outcome: Mean Change From Baseline in Composite Scores, National Eye Institute Visual Functioning Questionnaire (NEI-VFQ-25) at Months 3, 12 and 24
Description: The National Eye Institute Visual Function Questionnaire-25 (NEI-VFQ-25) was used to measure a patient's subjective assessment of vision-related quality of life at Months 3, 12 and 24. The 12 subscales in the VFQ-25 are general health, general vision, ocular pain, near activities, distance activities, social function, mental health, role difficulties, dependency, driving, color vision, and peripheral vision. The scores on the subscales were added together for a total score, which ranged from 0 to 100. A higher score indicated poorer function.
Time Frame: Baseline, Month 3, Month 12, Month 24
Population: All patients with a value for both baseline and the specific post-baseline visit. The baseline value is the last available, non-missing, value collected prior to first study treatment in the study eye.
Measure: Least Squares Mean (Standard Deviation); unit: Unit of scales
Arm/Group | Ranibizumab 0.5 mg + vPDT | Ranibizumab 0.5 mg | Ranibizumab 0.5 mg + vPDT (Switched)
Number analyzed (Participants) | 168 | 113 | 41
Unit of scales
  Month 3 - Value at Baseline: number analyzed (Participants) | 160 | 109 | 40
  Month 3 - Value at Baseline | 76.5 (13.78) | 75.9 (14.7) | 80.9 (12.47)
  Month 3 - Value at Visit | 79.4 (13.38) | 80.5 (12.21) | 82.5 (11.53)
  Month 3 - Change from Baseline | 2.9 (9.34) | 4.6 (10.52) | 1.7 (8.85)
  Month 12 - Value at Baseline: number analyzed (Participants) | 155 | 96 | 41
  Month 12 - Value at Baseline | 76.4 (13.6) | 75.8 (15.2) | 80.3 (12.77)
  Month 12 - Value at Visit | 82.8 (13.55) | 81.2 (13.54) | 83 (11.18)
  Month 12 - Change from Baseline | 6.4 (12.31) | 5.4 (13.54) | 2.7 (13.76)
  Month 24 - Value at Baseline: number analyzed (Participants) | 146 | 87 | 41
  Month 24 - Value at Baseline | 76.4 (13.72) | 76 (15.48) | 80.3 (12.77)
  Month 24 - Value at Visit | 81.9 (14.12) | 80.8 (13.37) | 83.2 (12.12)
  Month 24 - Change from Baseline | 5.5 (13.23) | 4.8 (14.92) | 2.8 (15.69)

17. Secondary Outcome: Number of Ocular Adverse Events of the Study Eye Regardless of Study Drug Relationship up to Month 24, Any Primary System Organ Class
Description: Reported categorically: Mild, Moderate, Severe
Time Frame: Up to Month 24
Population: Safety Analysis Set
Measure: Number; unit: Adverse Events
Arm/Group | Ranibizumab 0.5 mg + vPDT | Ranibizumab 0.5 mg | Ranibizumab 0.5 mg + vPDT (Switched)
Number analyzed (Participants) | 172 | 135 | 14
Adverse Events
  Mild | 55 | 31 | 7
  Moderate | 7 | 11 | 1
  Severe | 2 | 7 | 0

18. Secondary Outcome: Number of Non-Ocular Adverse Events of the Study Eye Regardless of Study Drug Relationship up to Month 24, Any Primary System Organ Class
Description: Reported categorically: Mild, Moderate, Severe
Time Frame: Up to Month 24
Population: Safety Analysis Set
Measure: Number; unit: Adverse Events
Arm/Group | Ranibizumab 0.5 mg + vPDT | Ranibizumab 0.5 mg | Ranibizumab 0.5 mg + vPDT (Switched)
Number analyzed (Participants) | 172 | 135 | 14
Adverse Events
  Mild | 65 | 49 | 6
  Moderate | 17 | 17 | 2
  Severe | 12 | 6 | 1

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) are collected from First Patient First Visit (FPFV) until Last Patient Last Visit (LPLV). All AEs reported in this record are from date of First Patient First Treatment until Last Patient Last Visit.
Description: All safety evaluations were carried out on the Safety set. The Safety Set consisted of all patients who received at least one application of study drugs and had at least one post-baseline safety assessment. The statement that a patient had no AEs also constituted a safety assessment. Within the safety set, patients were analyzed as treated.
Groups:
- Ranibizumab 0.5 mg + vPDT (Switched): Ranibizumab 0.5 mg + vPDT (Switched)
Arm/Group | Ranibizumab 0.5 mg + vPDT | Ranibizumab 0.5 mg | Ranibizumab 0.5 mg + vPDT (Switched)
All-Cause Mortality (participants affected / at risk) | 2/172 | 1/135 | 0/14
Serious Adverse Events (participants affected / at risk) | 27/172 | 23/135 | 2/14
Other Adverse Events (participants affected / at risk) | 80/172 | 45/135 | 11/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ranibizumab 0.5 mg + vPDT (N=172) | Ranibizumab 0.5 mg (N=135) | Ranibizumab 0.5 mg + vPDT (Switched) (N=14)
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 0
Anaemia of chronic disease (Blood and lymphatic system disorders) | 0 | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 1 | 0
Cardiac valve disease (Cardiac disorders) | 0 | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 1 | 0
Blindness unilateral (Study eye) (Eye disorders) | 0 | 1 | 0
Cataract (Fellow untreated eye) (Eye disorders) | 2 | 0 | 0
Cataract (Study eye) (Eye disorders) | 1 | 0 | 0
Macular hole (Study eye) (Eye disorders) | 1 | 0 | 0
Ocular hypertension (Study eye) (Eye disorders) | 0 | 1 | 0
Polypoidal choroidal vasculopathy (Fellow untreated eye) (Eye disorders) | 1 | 0 | 0
Retinal haemorrhage (Study eye) (Eye disorders) | 0 | 1 | 0
Vitreous haemorrhage (Fellow treated eye) (Eye disorders) | 0 | 1 | 0
Vitreous haemorrhage (Study eye) (Eye disorders) | 1 | 3 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 2 | 0 | 0
Campylobacter colitis (Infections and infestations) | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 1 | 0
Endophthalmitis (Study eye) (Infections and infestations) | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1 | 1
Pneumonia (Infections and infestations) | 1 | 4 | 0
Pneumonia bacterial (Infections and infestations) | 1 | 0 | 0
Wound infection (Infections and infestations) | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 2 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 2 | 0
Heat exhaustion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0
Embolic stroke (Nervous system disorders) | 0 | 1 | 0
Haemorrhagic stroke (Nervous system disorders) | 1 | 0 | 0
Presyncope (Nervous system disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Vocal cord leukoplakia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Aortic dissection (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ranibizumab 0.5 mg + vPDT (N=172) | Ranibizumab 0.5 mg (N=135) | Ranibizumab 0.5 mg + vPDT (Switched) (N=14)
Cerumen impaction (Ear and labyrinth disorders) | 0 | 0 | 2
Corneal disorder (Fellow untreated eye) (Eye disorders) | 0 | 0 | 1
Corneal disorder (Study eye) (Eye disorders) | 0 | 0 | 1
Dry eye (Fellow untreated eye) (Eye disorders) | 9 | 4 | 1
Dry eye (Study eye) (Eye disorders) | 10 | 4 | 1
Dyschromatopsia (Study eye) (Eye disorders) | 0 | 1 | 1
Eye irritation (Study eye) (Eye disorders) | 1 | 0 | 1
Lacrimation increased (Study eye) (Eye disorders) | 1 | 1 | 1
Ocular hyperaemia (Fellow untreated eye) (Eye disorders) | 0 | 0 | 1
Ocular hyperaemia (Study eye) (Eye disorders) | 1 | 0 | 1
Ocular hypertension (Study eye) (Eye disorders) | 3 | 3 | 1
Punctate keratitis (Fellow untreated eye) (Eye disorders) | 0 | 0 | 1
Punctate keratitis (Study eye) (Eye disorders) | 1 | 3 | 1
Retinal haemorrhage (Study eye) (Eye disorders) | 12 | 4 | 1
Retinal vein occlusion (Fellow untreated eye) (Eye disorders) | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 5 | 2 | 1
Dental caries (Gastrointestinal disorders) | 3 | 2 | 1
Gastritis erosive (Gastrointestinal disorders) | 0 | 0 | 1
Injection site pain (Study eye) (General disorders) | 1 | 0 | 1
Mass (General disorders) | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 23 | 10 | 2
Periodontitis (Infections and infestations) | 1 | 1 | 1
Pharyngitis (Infections and infestations) | 3 | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 0 | 1
Rhinitis (Infections and infestations) | 0 | 1 | 1
Tonsillitis (Infections and infestations) | 1 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 12 | 2 | 2
Foreign body in eye (Fellow untreated eye) (Injury, poisoning and procedural complications) | 0 | 0 | 1
Foreign body in eye (Study eye) (Injury, poisoning and procedural complications) | 0 | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 1
Intraocular pressure increased (Investigations) | 0 | 0 | 1
Intraocular pressure increased (Study eye) (Investigations) | 11 | 3 | 4
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 0 | 1
Fasciitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 4 | 1
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 6 | 5 | 1
Headache (Nervous system disorders) | 3 | 3 | 1
Visual field defect (Study eye) (Nervous system disorders) | 2 | 0 | 1
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 4 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 2 | 1 | 1
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 3 | 1 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 3 | 1 | 1
Hypertension (Vascular disorders) | 4 | 5 | 1
Varicose vein (Vascular disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.